CLINICAL TRIAL: NCT04906551
Title: Measuring Endometrial Blood Flow Using Laser Doppler: Acceptability & Reproducibility
Acronym: EMBeD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mary Eyo, Chief Investigator, Birmingham Women's and Children's NHS Foundation Trust
Other Study IDs: 250444
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Endometrium; Vascularization
MeSH Terms: conditions — Neovascularization, Pathologic | interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: laser Doppler — A direct measure of blood flow

SUMMARY:
35 participants will be recruited from a list of patients who are scheduled, as part of their routine NHS care, to have a clinically-indicated outpatient hysteroscopy for assessment of their uterine cavity. The participants will be women from the age of 18 up to the age of 40 who are undergoing hysteroscopy investigation. All participants included in the study require at least one ultrasound scan, within the preceding 5 years, demonstrating the presence of a normal uterine cavity devoid of uterine anomalies such as a septate uterus or intrauterine fibroids (which may affect endometrial blood flow measurements). It is usual for a patients to have an ultrasound assessment prior to hysteroscopy therefore we do not anticipate this requirement limiting the number of eligible participants available.

DETAILED DESCRIPTION:
Patient registry: Recruited patients will be registered on 'Edge', a secure, password-protected, database for study participants.

All the investigators will comply with the requirements of the GDPR 2018 with regards to the storage, processing and disclosure of personal information and will uphold the Act's core principles.

Access to patient-identifiable data will be restricted to the core patient-facing members of the research team at Birmingham Women's and Children's Hospital. The patient-facing members will be the Chief Investigator (ME), the Principal Investigator (JC), and co-investigator (HH).

The study involves depersonalised data and the data will be maintained within secure servers. The Birmingham Women's Hospital Research and Development department will hold an archived copy of the study data.

The Chief Investigator (ME) and the Principal Investigator (JC) will act as data custodians and keep the site file locked away securely with restricted access to study data for 25 years. Only the aforementioned members of the research team will have access to the site file for the purpose of quality control, audit and analysis.

Coded, depersonalised data will be created and used for study documents, in place of participant-identifying information. The participant data within the study and the code linking this data to the individual's true identity and identifiable data will be kept in separate locations using encrypted digital files within password-protected folders and storage media

ELIGIBILITY:
Inclusion Criteria:

* Women from the age of 18 up to the age of 40 who have consented to hysteroscopy investigation as part of their standard NHS care.
* Women who have had an ultrasound scan, within the preceding 5 years, demonstrating a normal uterine cavity with no gross anatomical abnormalities (e.g. uterine septum).
* Women who have given informed consented to take part in the study

Exclusion Criteria:

* Inability to tolerate vaginal examinations
* Women who are pregnant
* Women who do not have regular menstrual cycles
* Women who have not given consent to the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women from the age of 18 up to the age of 40 who have consented to hysteroscopy investigation as part of their standard NHS care.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-06-06 (Estimated); Study Completion 2022-06-06 (Estimated)

PRIMARY OUTCOMES:
The intra-operator variability | 1 minute
  The intra-operator variability of the 3 endometrial blood flow values taken for each participant, by a given operator.
The inter-operator variability | 1 minute
  The inter-operator variability, standard deviation, standard error and the variability of measurements taken between participants.

SECONDARY OUTCOMES:
Participant acceptability | 5 minutes
  Participant acceptability of undergoing laser Doppler measurement of endometrial tissue blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Mary Eyo, Principal Investigator — Birmingham Women's NHS Foundation Trust
Locations (1):
- BWC, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No